CLINICAL TRIAL: NCT01683123
Title: Phase 2 Study With Intravenous Busulfan And Fludarabine Myeloablative Conditioning For HLA Identical Sibling Allogeneic HSCT In Myeloid Malignancies. Retrospective Analysis.
Brief Title: Study With Intravenous Busulfan And Fludarabine Myeloablative Conditioning Regimen For HLA Identical Sibling Donor HSCT
Acronym: BUFLU
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Other Study IDs: get-buf-2010-02
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Myeloproliferative Disorders; Chronic Myeloid Leukemia
Keywords: Allogeneic HSCT; Busulfan; Fludarabina
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Analyze the results of conditioning with once-daily dose intravenous busulfan and fludarabine in patients undergoing HLA identical sibling Allogeneic HSCT for myeloid malignancies.

DETAILED DESCRIPTION:
In this study the investigators evaluate a conditioning regimen consisting in Fludarabine 40 mg/m2 once daily i.v in 60 min. on days -6 to -3 (total dose 160 mg/m2), followed by Busulfan 3,2 mg/kg once daily i.v. in 180 min. in the same days (total dose 12,8 mg/kg). No busulfan pharmacokinetic monitoring is performed. Graft versus host disease prophylaxis consists in the combination of cyclosporine and methotrexate. Graft products obtained from bone marrow or peripheral blood of HLA identical sibling donors are not manipulated in their cellular content before transplantation. Blood products were leukocyte depleted and irradiated before transfusion. Supportive care, including seizure prophylaxis, isolation measures, antiemetics, antimicrobial agents and growth factors use are followed according to standard procedures.

The main objectives are to record data regarding engraftment, regimen related toxicity and outcome in different patient populations according to age, disease type, disease status at HSCT and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myeloid Leukemia
* Myelodysplastic Syndrome
* Myeloproliferative Disorders
* Chronic Myeloid Leukemia

Exclusion Criteria:

* Performance status ECOG>2
* Cardiomyopathy (LVEF <39%)
* Pulmonary dysfunction (DLCO<39%)
* Hepatic dysfunction Grade >1
* Renal dysfunction Grade >1 (Creatinine > 1.6 mg/dl)
* HIV infection
* Other active neoplasm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with myeloid malignancies submitted to allogeneic HSCT with an HLA identical sibling donor
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier De la Serna, MD, Principal Investigator — Grupo Espanol de trasplantes hematopoyeticos y terapia celular; Guillermo Sanz, MD, Study Chair — Grupo Espanol de trasplantes hematopoyeticos y terapia celular